CLINICAL TRIAL: NCT02960581
Title: A Phase 1 Randomized Placebo-controlled Clinical Trial of the Safety, Pharmacokinetics and Antiviral Activity of PGT121 Monoclonal Antibody (mAb) in HIV-uninfected and HIV-infected Adults
Brief Title: Safety, PK and Antiviral Activity of PGT121 Monoclonal Antibody in HIV-uninfected and HIV-infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Beth Israel Deaconess Medical Center, Boston MA (Unknown); Ragon Institute of MGH, MIT and Harvard, Boston MA (Unknown); University of Texas Health, Houston AIDS Research Team (HART), Houston TX (Unknown); Mills Clinical Research, Los Angeles CA (Unknown); Orlando Immunology Clinic, Orlando FL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAVI T001
Record Dates: First submitted 2016-10-18; First posted 2016-11-09 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- Group 1A (Experimental): HIV-uninfected participants
  Interventions: Biological: PGT121 3mg/kg IV; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
- Group 1B (Experimental): HIV-uninfected participants
  Interventions: Biological: PGT121 10mg/kg IV; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
- Group 1C (Experimental): HIV-uninfected participants
  Interventions: Biological: PGT121 30mg/kg IV; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
- Group 2A (Experimental): HIV-infected on ART, (<50 cp/ml)
  Interventions: Biological: PGT121 3mg/kg IV; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
- Group 2B (Experimental): HIV-infected on ART, (<50 cp/ml)
  Interventions: Biological: PGT121 10mg/kg IV; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
- Group 2C (Experimental): HIV-infected on ART, (<50 cp/ml)
  Interventions: Biological: PGT121 30mg/kg IV; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
- Group 3A (Experimental): HIV-Infected off ART (VL 2x10^3 - 1x10^5 cp/ml)
  Interventions: Biological: PGT121 30mg/kg IV
- Group 3B (Experimental): HIV-Infected off ART (VL 1x10^2 - 2x10^3 cp/ml)
  Interventions: Biological: PGT121 30mg/kg IV
- Arm 1D (Experimental): HIV-uninfected participants
  Interventions: Biological: PGT121 3mg/kg SC; Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))

INTERVENTIONS:
Biological: PGT121 3mg/kg IV — 3mg/kg administered by IV Infusion
  Arms: Group 1A; Group 2A
Biological: PGT121 10mg/kg IV — 10mg/kg administered by IV infusion
  Arms: Group 1B; Group 2B
Biological: PGT121 30mg/kg IV — 30mg/kg administered by IV infusion
  Arms: Group 1C; Group 2C; Group 3A; Group 3B
Biological: PGT121 3mg/kg SC — 3mg/kg administered by SC injection
  Placebo: None
  Arms: Arm 1D
Biological: Placebo (0.9% Sodium Chloride Injection USP (Saline))
  Arms: Arm 1D; Group 1A; Group 1B; Group 1C; Group 2A; Group 2B; Group 2C

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, pharmacokinetics and anti-viral efficacy of the PGT121 monoclonal antibody for HIV prevention and therapy.

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the safety, tolerability, pharmacokinetics and anti-viral efficacy of the PGT121 monoclonal antibody for HIV prevention and therapy. PGT121 mAb is a recombinant human IgG1 monoclonal antibody that targets a V3 glycan-dependent epitope region of the HIV envelope protein. PGT121 mAb was chosen for this study because it is potent, neutralizes a wide array of HIV viruses, and can prevent and treat simian-human immunodeficiency virus (SHIV) in rhesus monkeys.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* HIV-uninfected males or females age 18-50 years old
* Willing to maintain low risk behavior for HIV infection

Group 1 Exclusion Criteria:

* confirmed HIV-infection, pregnancy or lactation, significant acute or chronic disease and clinically significant laboratory abnormalities

Group 2 Inclusion Criteria:

* HIV-infected males or females age 18-65 years old
* On a stable antiretroviral regimen with HIV-1 RNA plasma level <50 copies/ml, CD4 cell count greater than or equal to 300 cells/uL

Group 2 Exclusion Criteria:

* history of AIDS-defining illness within the previous 5 years, significant acute or chronic medical condition other than HIV infection, and clinically significant laboratory abnormalities

Group 3 Inclusion Criteria:

* HIV-infected males or females age 18-65
* Not on antiretroviral therapy for > 6 months with detectable HIV-1 viral load between 100 and 100,000 copies/ml, CD4 cell count greater than or equal to 300 cells/uL

Group 3 Exclusion Criteria:

* history of AIDS-defining illness within the previous 5 years, significant acute or chronic medical condition other than HIV infection, and clinically significant laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with PGT121 mAb reactogenicity, related AEs and SAEs | 6 Months post infusion
  The investigators will measure the following endpoints to evaluate the safety and tolerability of PGT121 mAb in HIV-uninfected and HIV-infected adults:
  1. Proportion of participants with moderate or greater reactogenicity (e.g., solicited adverse events) for 3 days following IV infusion of PGT121 mAb.
  2. Proportion of participants with moderate or greater and/or PGT121 mAb-related unsolicited adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, following IV infusion of PGT121 mAb for the first 56 days post administration of Investigational Product.
  3. Proportion of participants with PGT121 mAb-related serious adverse events (SAEs) throughout the study period.
Pharmacokinetics: elimination half-life (t1/2) | 6 Months post infusion
  Pharmacokinetics: elimination half-life (t1/2)
Pharmacokinetics: Clearance (CL/F) | 6 Months post infusion
  Pharmacokinetics: Clearance (CL/F)
Pharmacokinetics: Volume of distribution (Vz/F) | 6 months post infusion
  Pharmacokinetics: Volume of distribution (Vz/F)
Pharmacokinetics: Area under the concentration decay curve (AUC) | 6 months post infusion
  Pharmacokinetics: Area under the concentration decay curve (AUC)
Pharmacokinetics: Impact of viral load and/or ART on PGT121 disposition, volume of distribution, total exposure | 6 months post infusion
  Pharmacokinetics: Impact of viral load and/or ART on PGT121 disposition, volume of distribution, total exposure
Antiviral Activity | 6 Months post infusion
  Change in plasma HIV-1 RNA levels from baseline (mean of pre-entry and entry values)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Stephenson, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center, Center for Virology and Vaccine Research; Boris Juelg, MD PhD, Study Chair — Ragon Institute
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Stephenson KE, Julg B, Tan CS, Zash R, Walsh SR, Rolle CP, Monczor AN, Lupo S, Gelderblom HC, Ansel JL, Kanjilal DG, Maxfield LF, Nkolola J, Borducchi EN, Abbink P, Liu J, Peter L, Chandrashekar A, Nityanandam R, Lin Z, Setaro A, Sapiente J, Chen Z, Sunner L, Cassidy T, Bennett C, Sato A, Mayer B, Perelson AS, deCamp A, Priddy FH, Wagh K, Giorgi EE, Yates NL, Arduino RC, DeJesus E, Tomaras GD, Seaman MS, Korber B, Barouch DH. Safety, pharmacokinetics and antiviral activity of PGT121, a broadly neutralizing monoclonal antibody against HIV-1: a randomized, placebo-controlled, phase 1 clinical trial. Nat Med. 2021 Oct;27(10):1718-1724. doi: 10.1038/s41591-021-01509-0. Epub 2021 Oct 7. PMID 34621054
- See also: International AIDS Vaccine Initiative — http://iavi.org